CLINICAL TRIAL: NCT02956668
Title: tDCS Associated to Blindsight Rehabilitation for the Treatment of Homonymous Hemianopsia
Acronym: TABRTHH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 264-BSTDCS
Record Dates: First submitted 2016-10-27; First posted 2016-11-07 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Hemianopsia
Keywords: tDCS; Visual field; Stroke
MeSH Terms: conditions — Hemianopsia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blindsight training associated to tDCS (Experimental): During the blindsight training (one-hour time), the patient is asked to maintain central fixation and is exposed to visual stimuli in his blind hemifield. The patient task is detection and/or discrimination of stimuli.
  During each session the patient is subjected to around 700 different stimuli variously associated in space and/or time.
  tDCS stimulation start at the beginning of the rehabilitation session, and continue for 30 min, during treatment.
  Anode is placed over the parieto-occipital cortex. The cathode is placed in the contralateral supraorbital position.
  Interventions: Other: Blindsight Training associated to tDCS
- Blindsight training alone (Active Comparator): During the blindsight training (one-hour time), the patient is asked to maintain central fixation and is exposed to visual stimuli in his blind hemifield. The patient task is detection and/or discrimination of stimuli.
  During each session the patient is subjected to around 700 different stimuli variously associated in space and/or time.
  Interventions: Other: Blindsight Training alone

INTERVENTIONS:
Other: Blindsight Training associated to tDCS — The patient undergo visual rehabilitation while his brain is electrically stimulated with tDCS.
  Arms: Blindsight training associated to tDCS
Other: Blindsight Training alone — The patient undergo visual rehabilitation
  Arms: Blindsight training alone

SUMMARY:
Homonymous hemianopia is one of the most common symptoms following a neurologic damage and has many negative effects on functional abilities and daily activities.

There are two main kind of restorative rehabilitation of hemianopia: "border training", which involves exercising vision at the edge of the damaged visual field, and "blindsight training", which is based on exercising the unconscious perceptual functions in the mild of the blind hemifield.

In literature only border training effects were shown to be facilitated by transcranial direct current stimulation (tDCS).

The investigators treat two patients with blindsight rehabilitation associated to tDCS over parieto-occipital cortex. The two patients undergo a cycle of blindsight treatment associated to tDCS and a cycle of blindsight training alone in inverted order.

Aim of the study is to investigate if the anodic stimulation of perilesional areas enhance the improvement induced by blindsight rehabilitation treatment.

DETAILED DESCRIPTION:
The study design is a crossover AB BA. Treatment A consist in a cycle of blindsight training associated to tDCS, Treatment B consist in a a cycle of blindsight training alone.

During the blindsight training, the patient is asked to maintain central fixation and is exposed to visual stimuli in his blind hemifield. The patient task is detection and/or discrimination of stimuli.

During each session the patient is subjected to around 700 different stimuli variously associated in space and/or time.

One out of two blindsight training cycles is associated to tDCS treatment. Anodal tDCS is applied using a battery-driven constant current stimulator, and a pair of surface saline-soaked sponge electrodes (5 x 5 cm). Current intensity is of 2 mA (Fade-in/-out= 10 sec), for a total duration of 30 min. The stimulation start at the beginning of the rehabilitation session, and continue for 30 min, during treatment.

Anode is placed over the parieto-occipital cortex. The cathode is placed in the contralateral supraorbital position.

To assess the actual improvement patients performed:

1. Clinical-instrumental assessment: Threshold visual field Humphrey SITA-standard 30-2 program is used to measure the visual perception within the central 30 degrees.
2. Peripheral visual field test Schofield Vienna PP-R test is used to measure the visual perception up to 180 degrees. A double task in central vision was performed in order to verify test reliability.
3. Functional visual field assessment: Test for Attention Performance (TAP - v. 2.3) visual field 92 stimuli subtest (26) is performed.
4. Ecological assessment: during initial and final interview an ICF profile of the subject is edited. The profile includes mainly the Activity and Participation categories of ICF.

All these investigations is performed before the treatment and after each cycle

ELIGIBILITY:
Inclusion Criteria:

* The subject is able to give his informed consent
* Stroke
* Hemianopsia brain damage documented by means of TAC or RMN
* Hemianopsia diagnosed by means automated visual field and Neurological Evaluation
* Time from lesion at least six months
* normal or corrected-to-normal visual acuity

Exclusion Criteria:

* Presence of Ophthalmologic neuropsychologic or psychiatric pathology
* Global cognitive deficit,
* Presence of other neurological pathology
* Presence of cardiac peacemaker
* Presence metallic or electronic items in the head or in the body
* Story/familiarity of epilepsy, taking medications that can induce epileptic crisis
* Severe heart disease
* History of high alcohol consumption
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Humphrey visual field 30.2 SITA standard test | 10 weeks and 20 weeks

SECONDARY OUTCOMES:
Change in Battery for Attentional Performance (TAP) subtest: Visual Field | 10 weeks and 20 weeks
International Classification of Functioning (ICF) | 20 weeks
Change in Schuhfried Vienna Test Peripheral Perception (PP-R) | 10 weeks and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara M Matteo, Principal Investigator — Università degli Studi di Milano - Bicocca
Locations (1):
- Polo universitario presso I.C. Zucchi, Carate Brianza, CB, Italy

IPD SHARING:
Plan to Share IPD: Undecided